CLINICAL TRIAL: NCT00888576
Title: A Registry Study to Describe the Implications of Therapeutic Management of Etanercept in Patients With Rheumatoid Arthritis
Brief Title: Registry of Etanercept Use in Patients With Rheumatoid Arthritis in Clinical Practice in Taiwan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-4445
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Non-intervention

SUMMARY:
The purpose of this study is to develop a registry with safety and efficacy data on the use of etanercept in clinical practice in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria: 1) Male or female patients aged > 20 years; 2) Patients who have already been selected and approved under the Taiwan National Health Insurance Program to receive 24 weeks of etanercept for rheumatoid arthritis. Main

Exclusion Criteria:

Exclusion Criteria: None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinic
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety: Proportion of patients discontinued from etanercept as a result of an adverse event by Week 24, laboratory exam findings, incidence of adverse events, and vital signs and physical exam findings. Efficacy: Disease Activity Score 28 at week 20. | 24 weeks

SECONDARY OUTCOMES:
Global health assessment; Erythrocyte sedimentation rate; Number of swollen or tender joints; C-reactive protein; Proportion of patients having worsened DAS 28 and components of DAS 28,CRP than baseline; Etanercept approval-lag time. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Taiwan (18):
  - Pfizer Investigational Site, Changhua, Changhua County
  - Pfizer Investigational Site, Changhua, Changhua
  - Pfizer Investigational Site, Lukang Zhen, Changhua
  - Pfizer Investigational Site, Dalin, Chia-Yi
  - Pfizer Investigational Site, Putz, Chiayi
  - Pfizer Investigational Site, Kaohsiung City, Kaohsiung
  - Pfizer Investigational Site, Niao Sung Hsiang, Kaohsiung
  - Pfizer Investigational Site, Keelung, Keelung
  - Pfizer Investigational Site, Taichung, Taichung
  - Pfizer Investigational Site, Taipei, Taipei
  - Pfizer Investigational Site, Taipei TOC, Taiwan
  - Pfizer Investigational Site, Guishanli, Taoyuan
  - Pfizer Investigational Site, Taoyuan District, Taoyuan
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4445&StudyName=Registry%20of%20etanercept%20use%20in%20patients%20with%20rheumatoid%20arthritis%20in%20clinical%20practice%20in%20Taiwan